CLINICAL TRIAL: NCT02049190
Title: A Phase 1-2 Study of Onapristone in Patients With Advanced Castration-resistant Prostate Cancer
Brief Title: Phase 1-2 Study of Onapristone in Patients With Advanced Castration-resistant Prostate Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arno Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARN-AR18-CT-102
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Prostate Cancer; Metastatic Prostate Cancer; Androgen-independent Prostate Cancer; Recurrent Prostate Cancer
Keywords: Advanced Prostate Cancer; Castration-resistant Prostate Cancer; Prostatic Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms; Neoplasms by Site; Neoplasms; Genital Diseases, Male; Prostatic Diseases; onapristone
MeSH Terms: conditions — Prostatic Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms; Neoplasms by Site; Neoplasms; Genital Diseases, Male; Prostatic Diseases | interventions — onapristone; abiraterone; Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- onapristone 10 mg BID (Experimental): onapristone 10 mg BID extended-release tablets
  Interventions: Drug: onapristone
- onapristone 20 mg BID (Experimental): onapristone 20 mg BID extended-release tablets
  Interventions: Drug: onapristone
- onapristone 30 mg BID (Experimental): onapristone 30 mg BID extended-release tablets
  Interventions: Drug: onapristone
- onapristone 40 mg BID (Experimental): onapristone 40 mg BID extended-release tablets
  Interventions: Drug: onapristone
- onapristone 50 mg BID (Experimental): onapristone 50 mg BID extended-release
  Interventions: Drug: onapristone
- onapristone 30 mg BID + abiraterone 1000 mg (Experimental): Expansion cohort: onapristone 30 mg BID + abiraterone 1000 mg
  Interventions: Drug: onapristone; Drug: abiraterone
- onapristone 50 mg BID + abiraterone 1000 mg (Experimental): Expansion cohort: onapristone 50 mg BID + abiraterone 1000 mg
  Interventions: Drug: onapristone; Drug: abiraterone
- Expansion cohort: onapristone 50 mg BID (Experimental): Expansion cohort: onapristone 50 mg BID
  Interventions: Drug: onapristone

INTERVENTIONS:
Drug: onapristone
  Other Names: ZK 98299
Drug: abiraterone
  Other Names: Zytiga
  Arms: onapristone 30 mg BID + abiraterone 1000 mg; onapristone 50 mg BID + abiraterone 1000 mg

SUMMARY:
This is an open-label, randomized, parallel group two-stage phase 1-2 study with an escalation and an expansion component. This study will evaluate an extended-release (ER) formulation of onapristone in patients with prostate cancer in which Progesterone Receptor (PR) may be contributing to tumor progression. A companion diagnostic to select patients whose prostate cancer expresses the activated form of the PR (APR) is under development and will be implemented in this study; it may be used to further enrich the selection of the population based upon ongoing review of the results. Patients will be treated until occurrence of an intolerable safety issue, treatment failure, if patient elects to withdraw, or for non-compliance with either protocol-specified evaluations or onapristone treatment. An additional cohort of patients will be included at the recommended phase 2 dose to gain additional understanding of the onapristone safety profile and potential anti-cancer activity.

ELIGIBILITY:
Inclusion criteria:

1. Male patients, 18 years of age or greater;
2. Histologically confirmed adenocarcinoma of the prostate (without neuroendocrine differentiation or small cell features);
3. In Stage 2, a mandatory biopsy is required with confirmed PR or APR in ≥1% tumor cells. For patients recruited to the abiraterone-onapristone combination arm, the biopsy must be performed on abiraterone administered as the most recent treatment and after a minimum of 2 weeks continuous treatment. For other patients, the biopsy must be taken at progression on or after abiraterone or enzalutamide or before screening with no anti-cancer treatment taken in the intervening period and a maximum of six (6) months prior to study start. If archival tissue is also available this should be provided for comparison purposes; a paired biopsy at day 8-28 is optional;
4. Metastatic or recurrent inoperable disease after previous surgery, radiation therapy, and/or chemotherapy;
5. For patients in Stage 1 and for patients in Stage 2 who will receive combination therapy with onapristone and abiraterone: no more than one prior chemotherapy regimen for CRPC (docetaxel rechallenge will be regarded as one line of chemotherapy); for patients in Stage 2 who will receive onapristone monotherapy: no prior chemotherapy is allowed;
6. Disease that has progressed by PSA or radiologically, on abiraterone or enzalutamide. Disease progression for study entry is defined as one or both of:

   * PSA progression defined by a minimum of two rising PSA levels with an interval of ≥1 week between each determination.
   * Radiological progression per RECIST 1.1;
7. For patients recruited to the abiraterone-onapristone combination arm, progression on abiraterone as their last line of treatment is required after a prior response to abiraterone;
8. The PSA value at screening and baseline should be ≥ 2 µg/L (2 ng/mL);
9. For onapristone monotherapy, corticosteroid discontinuation >4 weeks or >2 weeks with normal adrenal function confirmed by an ACTH stimulation test. For the combination onapristone - abiraterone arm, prednisolone 5mg BID and no other steroid regimen allowed for 2 weeks prior to treatment initiation;
10. Ongoing androgen deprivation therapy with a gonadotropin releasing hormone (GnRH) analogue or orchiectomy (i.e., surgical or medical castration);

    • For patients who have not had an orchiectomy, there must be a plan to maintain effective GnRH-analogue therapy for the duration of the trial;
11. Serum testosterone level < 1.7 nmol/L (50 ng/dL);
12. Patients receiving bisphosphonate therapy must have been on stable doses for at least 4 weeks;
13. Evaluable disease per RECIST 1.1 [Eisenhauer 2009] or Prostate Cancer Clinical Trials Working Group 2 (PCWG2) [Scher 2008];
14. ECOG performance status 0-2;
15. Life expectancy ≥ 3 months;
16. Willing and able to sign written informed consent per ICH-GCP, the local regulatory requirements, and local data protection laws prior to study-specific screening procedures.

Exclusion criteria:

1. Serum creatinine >1.5 ULN;
2. On ECG a QTc(F) interval >480 msec or any clinically significant cardiac rhythm abnormalities;
3. Liver function tests documented within the screening period and/or at baseline:

   1. Total bilirubin > ULN (except in patients diagnosed with Gilbert's disease);
   2. Alkaline phosphatase > 2.5 x UNL, unless test for alkaline phosphatase isoenzymes is elevated only for bone isoenzyme;
   3. ALT/AST > UNL or > 2.5 x UNL in case of liver metastases;
4. Absolute neutrophil count < 1,500/µL, platelet count < 100,000/µL, and hemoglobin < 5.6 mmol/L (9 g/dL) and no growth factors or blood transfusions within 7 days of these values;
5. Serum albumin < 25 g/L (2.5 g/dL);
6. Known positive virology/serology for human immunodeficiency virus (HIV)-1, HIV-2, hepatitis B (surface antigen), or hepatitis C (testing not required);
7. Chronic inflammatory liver condition. History or clinical evidence of any liver or biliary pathology including cirrhosis, infectious disease, inflammatory conditions, steatosis, or cholangitis (including ascending cholangitis, primary sclerosing cholangitis, obstruction, perforation, fistula of biliary tract, spasm of sphincter of Oddi, biliary cyst or biliary atresia;
8. Patients with any other prior malignancy are not allowed except for:

   1. Adequately treated basal cell or squamous cell skin cancer;
   2. Adequately treated Stage I or II cancer from which the patient is currently in complete remission;
   3. Other cancer from which the patient has been disease-free for 2 years;
9. For Stage 1 only: Chronic adrenal failure or is receiving concurrent long-term corticosteroid therapy. Prior long-term corticosteroids must be stopped ≥4 weeks or >2 weeks if normal adrenal function is confirmed by an ACTH stimulation test prior to start of study drug;
10. History or clinical evidence of any surgical or medical condition which the investigator judges as likely to interfere with the results of the study or pose an additional risk in participating; e.g., active or clinically significant history of disease involving a major organ system-vascular, cardiac, uncontrolled hypertension, pulmonary, gastrointestinal, hematologic, neurologic, neoplastic, renal, endocrine or immunodeficiency, or clinically significant active psychiatric disorders;
11. Used any prescription medication during the prior 2 weeks that the investigator judges is likely to interfere with the study or to pose an additional risk to the patient in participating, specifically inhibitors or inducers of cytochrome P450 (CYP)3A4 (see Appendix 4);
12. Received an investigational product or been treated with an investigational device within 30 days prior to first drug administration, or plans to start any other investigational product or device study within 30 days after last drug administration;
13. Received prior therapies within the following time period prior to receipt of first dose of study drug (Day 1, without withdrawal response and with no plans to initiate any of these during study:

    1. Ketoconazole or bicalutamide within 6 weeks;
    2. Systemic hormone therapy, chemotherapy, targeted therapies, antibodies within 4 weeks excluding abiraterone in the abiraterone-onapristone combination arm;
    3. Fractionated radiotherapy within 3 weeks;
    4. Single fraction of radiotherapy within 2 weeks;
    5. Radionuclide therapy within 8 weeks;
    6. Brachytherapy Pd-103 implant within the last 3 months;
    7. Brachytherapy I-125 implants within 12 months.
14. Concurrent use of herbal products that may decrease PSA levels (e.g., saw palmetto);
15. Residual toxicity of prior anticancer treatment > grade 1 except for alopecia;
16. Brain metastases, active epidural disease or spinal cord compression, unless treated at least 4 weeks before entry, and stable with steroid treatment for ≥1 week;
17. Paget's disease of the bone;
18. Structurally unstable bone lesions suggesting impending fracture;
19. Patients with reproductive potential not employing adequate contraception during treatment and for 1 month after completing treatment;
20. Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to swallow pills;
21. Mental incapacity or language barriers precluding adequate understanding, co-operation, and compliance with the study requirements;
22. Is, in the judgment of the investigator, unable or unwilling to comply with the requirements of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2014-02; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities related to onapristone or the combination of onapristone and abiraterone utilizing a day 57 safety cut off and based on CTCAE v4 | Baseline to 57 days post-first dose
Response to onapristone or the combination of onapristone and abiraterone | Baseline to 30 Days after last dose
  * Objective partial or complete response by RECIST 1.1, confirmed on a second CT scan at least 4 weeks apart and / or
  * PSA decline of ≥ 50% (according to the PCWG2).

SECONDARY OUTCOMES:
Safety and tolerability of extended-release onapristone tablets BID | Baseline to 30 Days after last dose
  Safety will be assessed by physical exam, vital signs, monitoring of adverse events, changes in ECG, and changes in PSA and other clinical laboratory values.
PK of onapristone, mono-demethylated onapristone and other metabolites in plasma and urine | Baseline to 30 Days after last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Inst of Cancer Research & Royal Marsden NHS Foundation Trust, Sutton Surrey, United Kingdom